CLINICAL TRIAL: NCT06944015
Title: Reduced-pressure Pneumoperitoneum and Intraperitoneal Saline Washout to Alleviate Pain Following vNOTES Hysterectomy
Acronym: Vnotes
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Erzincan Military Hospital (Other)
Responsible Party: Principal Investigator, Kemal GUNGORDUK, MD, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: M08; 250014/60 (Other: Mugla University)
Record Dates: First submitted 2025-04-17; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Pain, Inflammatory; Pain Management
MeSH Terms: conditions — Pain; Agnosia | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Saline (Experimental): After completion of VNOTE surgery, study Group patients underwent intraperitoneal irrigation with 30 mL/kg of normal saline at 37C infused under the right hemidiaphragm. Patients were placed in Trendelenburg position and reverse Trendelenburg position, to allow contact between the liquid and all abdominal structures, including the diaphragm. At the end of the procedure, the introduced liquid was carefully removed.
  Interventions: Other: normal saline
- Control Group (No Intervention): No intervention was performed after the vNOTES

INTERVENTIONS:
Other: normal saline — After completion of surgery, Study Group patients underwent intraperitoneal irrigation with 30 mL/kg of normal saline at 37C infused under the right hemidiaphragm. Patients were placed in Trendelenburg position and reverse Trendelenburg position, to allow contact between the liquid and all abdominal structures, including the diaphragm and surgical wounds. At the end of the procedure, all the introduced liquid was carefully removed.
  Arms: Normal Saline

SUMMARY:
vNOTES, initially employed for cholecystectomy, appendectomy, and nephrectomy, made its debut in the field of gynecologic surgery in 2012. The advantages of vNOTES-such as minimized postoperative discomfort, quicker recovery, and superior cosmetic results-combined with gynecologists' familiarity with the vaginal approach, have contributed to the swift global adoption of vNOTES in gynecological procedures. Preliminary trials have demonstrated its safety and practicality.

Although laparoscopy plays a crucial role in surgical procedures, post-operative pain remains a major concern linked to this minimally invasive technique, despite being less intense than the pain from a laparotomy. Visceral pain after laparoscopy can stem from the stretching of the peritoneum and diaphragm caused by pneumoperitoneum, as well as from inflammatory cytokines released due to blood accumulation in the abdominal cavity. This pain is typically described as a dull, widespread ache found in the abdominal or thoracic region and often extends to the shoulders. It corresponds to a rise in painkiller use aligned with Enhanced Recovery After Surgery strategies for both preoperative and postoperative stages. Moreover, the Trendelenburg position could intensify shoulder pain due to increased diaphragm irritation from pneumoperitoneum.

Effective pain management promotes early movement, lowering the risk of blood clots and decreasing lung complications like atelectasis or pneumonia. Additionally, postoperative pain negatively impacts the quality of life immediately after surgery. To lessen both the occurrence and intensity of post-surgical pain, numerous experts advocate for the use of multimodal therapy in surgical patients.

The aim of this study was to evaluate the efficacy of combined low-pressure CO2 pneumoperitoneum and intraperitoneal infusion of normal saline for reducing the incidence and severity of postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received vNOTES hysterectomy and salpingectomy, with the option of additional procedures such as oophorectomy, uterosacral ligament plications, transobturator tape insertion, colporrhaphy, or sentinel lymphadenectomy.
* ASA status I-III
* Voluntary participation

Exclusion Criteria:

* Surgery time greater than 3 h,
* suspected infection or malignancy or rectovaginal endometriosis
* participation in other clinical trials.
* presence of pre-surgical shoulder pain or any acute or chronic pain syndromes
* cognitive impairment or communications disorder,
* previous use of opioids for chronic pain,

Max Age: 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-04-24 (Estimated); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-03-16 (Estimated)

PRIMARY OUTCOMES:
the visual analogue scale (VAS) | 6 hours after surgery
  A Visual Analogue Scale (VAS) is an instrument for subjective rating of pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain (0)" and "worst pain (10)."

IPD SHARING:
Plan to Share IPD: No